CLINICAL TRIAL: NCT02829203
Title: Pre-Frailty Score as a Predictor Risk on Cardiovascular Surgery Outcome in Elderly
Brief Title: Pre-Frailty Risk in Cardiovascular Surgery
Status: Completed | Type: Observational
Sponsor: Instituto Dante Pazzanese de Cardiologia (Other)
Responsible Party: Principal Investigator, Mayron Faria de Oliveira, PhD, Instituto Dante Pazzanese de Cardiologia
Other Study IDs: 4560
Record Dates: First submitted 2016-07-04; First posted 2016-07-12 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Post Cardiac Surgery
Keywords: Frailty; Surgery
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- No-Frailty: Patients without frailty score submitted to a cardiac surgery
- Pre-Frailty: Patients with pre-frailty score submitted to a cardiac surgery

SUMMARY:
Frailty is an important risk factor for cardiovascular disease (CVD), recent data has shown significant association between pre-frailty and the risk of incident for CVD, irrespective of any classical cardiometabolic risk factors, suggesting that targeting pre-frailty as a potentially reversible risk factor for CVD in the elderly. Patients with high levels of frailty have an increased risk in post-operative period, with more time in mechanical ventilation, length of stay and complications (stroke and death) compared to patients with low frailty levels. The investigators hypothesized that pre-frailty patients also have a higher surgical risk compared to no-frailty patients.

DETAILED DESCRIPTION:
This was a prospective observational study involving patients over 65 years recruited from the Dante Pazzanese Institute of Cardiology. The patients had an established diagnosis of cardiovascular diseases (myocardial infarction or valve regurgitation) by previous electrocardiogram and/or Doppler echocardiography and all had surgical indication (coronary artery bypass, valve replacement or combined surgery). Patients with prior neurological disease (previous stroke or muscular dystrophies) or cognitive impairment resulting from previous injury or who refused to participate in the study were excluded.

Twenty-four hours before the surgery patients were evaluated by Frailty score as described elsewhere and divided into 2 groups: No-Frailty (Frailty score 1 or 2) and Pre-Frailty (Frailty score 3 or 4). If the patient had Frailty score higher than 5 were excluded from the study.

After surgery all patients were admitted at the intensive care unit (ICU) following the institutional mechanical ventilation protocol. Immediately after admission heart rate, mean arterial pressure, and oxygen pulse saturation (SpO2) were measured with a Dixtal monitor (DX 2010). After ICU admission all participants were followed up for main outcomes: hospital discharge, stroke, infection or death. In addition the investigators also measured length of stay, the duration of mechanical ventilation, vasopressors usage and the needed of physiotherapy indication after hospital discharge. All study participants receive medical and physiotherapy care according to the routine of the institution.

ELIGIBILITY:
Inclusion Criteria:

* cardiovascular diseases (myocardial infarction or valve regurgitation) by previous electrocardiogram and/or Doppler echocardiography and all had surgical indication (coronary artery bypass, valve replacement or combined surgery).

Exclusion Criteria:

* neurological disease (previous stroke or muscular dystrophies) or cognitive impairment resulting from previous injury or who refused to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients with an established diagnosis of cardiovascular diseases (myocardial infarction or valve regurgitation) by previous electrocardiogram and/or Doppler echocardiography and all had surgical indication (coronary artery bypass, valve replacement or combined surgery). Patients with prior neurological disease (previous stroke or muscular dystrophies) or cognitive impairment resulting from previous injury or who refused to participate in the study were excluded.
  Twenty-four hours before the surgery patients were evaluated by Frailty score as described elsewhere and divided into 2 groups: No-Frailty (Frailty score 1 or 2) and Pre-Frailty (Frailty score 3 or 4). If the patient had Frailty score ≥ 5 they were excluded from the study.
Sampling Method: Non-Probability Sample
Enrollment: 221 (Actual)
Dates: Start 2015-05; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Cardiac outcome in patients with or without frailty score | 6 months

IPD SHARING:
Plan to Share IPD: No